CLINICAL TRIAL: NCT03015870
Title: Technology-assisted Vocal Exercise for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB15130
Record Dates: First submitted 2015-11-04; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Aging
Keywords: vocal dysfunction; voice; vocal folds; vocal aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback (Experimental): Behavioral: Vocal exercise with real-time feedback.
  Interventions: Behavioral: Vocal exercise with real-time feedback
- Recording (Active Comparator): Behavioral: Vocal exercise with recording
  Interventions: Behavioral: Vocal exercise with recording

INTERVENTIONS:
Behavioral: Vocal exercise with real-time feedback — The feedback intervention will use iPads pre-installed with a PDF of vocal exercises for the full duration of the study and with an app which will provide tailored feedback regarding pitch, loudness, and duration of phonation during practice sessions.
  Arms: Feedback
Behavioral: Vocal exercise with recording — The recording intervention will use an iPad pre-installed with the PDF of vocal exercises for the full duration of the study, but no feedback app.Participants audio record self while performing vocal exercises
  Arms: Recording

SUMMARY:
Many detrimental effects of aging have been identified in the human voice, most of which are accepted as "normal". However, age-related vocal deficits disrupt communication and decrease quality of life in older adults and may be preventable and/or treatable through behavioral interventions. The objective of this proposal is to determine the effectiveness of a technology-assisted vocal exercise intervention on the vocal function and quality of life in older adults. Forty older adults (65+) will be recruited and randomly assigned to either an app or PDF-delivered vocal training intervention lasting 8 weeks. Pre- and post-testing involving vocal functioning assessments, as well as mobility, psychosocial, and cognitive functioning assessments will be conducted. This interdisciplinary project will enhance the investigators understanding of physical, mental, and social health-related quality of life among older adults.

DETAILED DESCRIPTION:
All participants will receive an iPad pre-loaded with an instructional PDF containing written instructions and embedded recorded audio prompts to assist with the delivery of an established vocal training paradigm, the Vocal Function Exercises (VFE) developed by Stemple.22 The VFE involves a set of four exercises focusing on extending maximum phonation time, increasing pitch range, and, therefore, improving coordination of the respiratory, phonatory, and resonatory systems during voicing. The iPads will be collected from the participants at the conclusion of the study at the post-intervention testing sessions.

Participants will be randomly assigned to either an experimental feedback group or active control no feedback group. Participants in the feedback group will receive iPads pre-loaded with Sonneta Voice Monitor app (MintLeaf Software) which will provide tailored feedback regarding pitch, loudness, and duration of phonation during practice sessions. The no feedback group will be provided with an iPad pre-installed with the PDF for the full duration of the study, but no feedback app.

Prior to and separate from the individual baseline testing appointments (described below), one group-based introductory session will be held to orient all participants to iPad controls (i.e., navigation, volume, recordings), as well as training specific to their assigned condition (how to use the pdf or app). Participants will complete a progressive weekly training schedule (3, 4, 5, 6, 7, 7, 7, & 7 days per week) 2x per day for 30-minute sessions over 8 weeks. The first training session will be monitored to provide technical assistance and ensure fidelity of the training protocol. Undergraduate research assistants from Dr. Johnson's lab will contact each participant via telephone on a weekly basis to provide technical assistance and confirm adherence to the training schedule.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Vision at least 20/40 with glass or contacts

Exclusion Criteria:

* Moderate-severe cognitive impairment
* Currently engaged in regular daily singing practice
* Currently involved in a research study involving exercise, memory, or vocal strengthening
* Currently being treated for a voice disorder by either an ENT or SLP

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Vocal acoustic function | 8-week change from baseline
  Dysphonia Severity Index: composite measure of maximum phonation time (s), highest fundamental frequency (Hz), lowest intensity (dB) and jitter (%).
Vocal aerodynamic function | 8-week change from baseline
  Phonation threshold pressure (kPa)

SECONDARY OUTCOMES:
Program engagement and app usability | 8-week training period
  Assessed via self-report (and verified via objective data) weekly during intervention and computed as an un-weighted composite score reflecting 8-week program adherence and ease of use.
Training-induced Change in Voice-related Quality of Life | 8-week change from baseline
  The London Chest Activity of Daily Living Scale will be used to assess theoretical and mechanistic components of the vocal exercise intervention. Un-weight composite scores will be calculated at each assessment.
Acceptability/feasibility of intervention | Post-intervention (8-week follow-up)
  Self-reported level of agreement (1 strongly disagree, 7 strongly agree) with three separate statements ("I enjoyed the program I used to exercise my voice," "I will continue to use the training techniques in the future," and "I believe my voice improved as a result of my participation in this program")
Respiratory Function | 8-week change from baseline
  FEV1 - forced expiratory volume in 1 second (Liters)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Johnson, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary data will be made available via https://databank.illinois.edu/ within 6 months of trial completion. Secondary data will be available within 2 years of trial completion.